CLINICAL TRIAL: NCT01046955
Title: Head-to-Head Comparison of Thymoglobulin vs. Campath-1H vs. Our Standard Center Treatment Protocol in Living Donor Renal Transplantation - A Study to Evaluate the Avoidance of Long-term Nephrotoxic Calcineurin Inhibitor Therapy
Brief Title: Thymoglobulin Versus Alemtuzumab Versus Daclizumab in Living Donor Renal Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: George Burke, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 20010704
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2008-05

CONDITIONS: End-Stage Renal Disease; Living Donors
Keywords: ESRD
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — thymoglobulin; Daclizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1mg/kg Thymoglobulin (Active Comparator): LD kidneys receiving 1mg/kg Thymoglobulin for 7 days starting at the day of surgery.
  Interventions: Drug: Anti-Thymocyte Globulin vs Campath-1H vs Daclizumab
- Campath-1H at 0.3 mg/kg (Active Comparator): Recipients of LD kidneys receiving Campath-1H at 0.3 mg/kg once on the day of surgery and again 3 days post-operatively.
  Interventions: Drug: Anti-Thymocyte Globulin vs Campath-1H vs Daclizumab
- Zenapax 1 mg/kg (Active Comparator): Recipients of LD kidneys receiving Zenapax 1mg/kg on the day of surgery followed by the same dose every 2 weeks for a total of 5 dosages.
  Interventions: Drug: Anti-Thymocyte Globulin vs Campath-1H vs Daclizumab

INTERVENTIONS:
Drug: Anti-Thymocyte Globulin vs Campath-1H vs Daclizumab — comparison of induction therapies.
  Other Names: Thymoglobulin; Zenapax

SUMMARY:
The purpose of this study is to observe in a randomized prospective study the effectiveness and toxicity of Thymoglobulin vs. Campath-1H used for induction therapy in recipients of living donor (LD) kidneys, compared with the investigators standard treatment protocol of Zenapax® and maintenance immunosuppression.

DETAILED DESCRIPTION:
To observe in a randomized prospective pilot study the effectiveness and toxicity of Thymoglobulin vs. Campath-1H used for induction therapy in recipients of living donor (LD) kidneys, compared with our standard treatment protocol of Zenapax® and maintenance immunosuppression (vide infra).

To determine the effect different antibody induction regimen on the lymphoid cell subsets of the immune system in kidney allograft recipients peripheral blood and bone marrow aspirates will be tested at surgery before transplantation and at intervals post operatively.

To treat renal transplant patients successfully in the absence of long-term calcineurin inhibition to determine if there are beneficial effects on the prevention of chronic allograft nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Age >14 years
* Weight >40 kg
* Primary renal allograft:living related (non HLA identical) and unrelated donor
* Negative standard cross match for T-cells
* Signed and dated consent form

Exclusion Criteria:

* Patient has previously received or is receiving an organ transplant other than kidney
* Patient has received a kidney transplant from a non-heart beating donor
* Patient has received an ABO incompatible donor kidney
* Recipient or donor is seropositive for human immunodeficiency virus (HIV)
* Patient has a current malignancy or a history of malignancy

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-11; Primary Completion 2007-04 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To observe in a randomized prospective pilot study the effectiveness and toxicity of Thymoglobulin vs. Campath-1H used for induction therapy in recipients of living donor kidneys. | 3 years
Patient/graft survival. | 1 and 3 yrs.

SECONDARY OUTCOMES:
Incidence of adverse reactions. | 1 & 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: George W Burke, M.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami Jackson Memorial Hospital, Miami, Florida, United States